CLINICAL TRIAL: NCT06036069
Title: Improvement of Whole Body Vibration and Core Stability Exercises on Muscle Strength in Down Syndrome Children
Brief Title: Effect of Whole Body Vibration Versus Core Stability Exercises on Balance and Muscle Strength in Children With Down Syndrome
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ragaee Saeed Mahmoud (Other)
Responsible Party: Sponsor-Investigator, Ragaee Saeed Mahmoud, Lecturer, South Valley University
Organization: South Valley University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P.T.REC/012/004335
Record Dates: First submitted 2023-09-02; First posted 2023-09-13 (Actual); Last update posted 2023-10-13 (Actual); Status verified 2023-10

CONDITIONS: Down Syndrome
Keywords: Children; Core Stability Exercises; Down Syndrome; Whole Body Vibration
MeSH Terms: conditions — Down Syndrome

STUDY DESIGN:
Intervention Model Description: Randomized control study
Who Masked: Outcomes Assessor
Masking Description: Single (outcomes Assessor)
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Conventional physical therapy group (Experimental): It consisted of 20 children received conventional physical therapy
  Interventions: Other: Conventional physical therapy
- Core stability exercises group (Experimental): It consisted of 20 children received conventional physical therapy and core stability exercises
  Interventions: Other: Conventional physical therapy
- Whole body vibration (Experimental): It consisted of 20 children received conventional physical therapy and whole body vibration exercises
  Interventions: Other: Conventional physical therapy

INTERVENTIONS:
Other: Conventional physical therapy — * Standing with feet together while the therapist was sitting behind and manually locking the child knees.
  * Step standing with the therapist behind the child.
  * High step standing and trying to keep balanced. The child stood on exercise mattress.
  * Single leg stance "unilateral standing" with assistance. The child was standing on exercise mattress.
  * Standing on a declined surface by using wedge. The child was standing on wedge towards the descending direction.
  * Standing with manual locking of the knees.
  * Changing position.
  * Gait training.
  * Static and dynamic muscle contraction.
  Other Names: Physical therapy program

SUMMARY:
Children had Down syndrome often have impaired balance and postural control and result as less active than their peers that can lead to reduced quality of life and movement skills. Effects of physical activity may be important in preventing falling risk and health consequences in those children

DETAILED DESCRIPTION:
Sixty children from both genders (boys and girls) participated in this study, their ages ranged from 10 to 16 years and they were randomized into three groups of same number (A, B and C). Groups (A) received conventional physical therapy program, group (B) received the same conventional physical therapy program of group (A) and core stability exercises while group (C) received the same conventional physical therapy program of group (A and B) and whole body vibration exercise

ELIGIBILITY:
Inclusion Criteria:

* Aged between 10 to 16 years.
* Able to recognize commands given to them.
* Understand our verbal command and encouragement.
* Stand and walk independently without repeated falling.

Exclusion Criteria:

* Children with any neurological (signs of epilepsy and instability of atlantoaxial joint).
* Musculoskeletal, or mobility disorders.
* Cardiac anomalies.
* Vision or hearing loss.

Ages: 10 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2023-10-15 (Estimated); Primary Completion 2024-01-15 (Estimated); Study Completion 2024-01-20 (Estimated)

PRIMARY OUTCOMES:
Biodex Balance System | before intervention and after 12 weeks of intervention
  it is a reliable and objective assessment in order to quantify dynamic balance

SECONDARY OUTCOMES:
Hand-held dynamometer | before intervention and after 12 weeks of intervention
  It is a portable device (Nicholas Manual Muscle Tester, Model 01160; Lafayette Instrument, Lafayette, IN), characterized as low-cost and convenient method

CONTACTS AND LOCATIONS:
Locations (1):
- Ragaee Saeed Mahmoud, Giza, Faisal, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol